CLINICAL TRIAL: NCT04467372
Title: The Effects Supplementation of Tart Cherry or Placebo on the Gut Microbiome, Inflammation, Oxidative Stress, and Health-related Outcomes.
Brief Title: Tart Cherry Supplementation & Gut Microbiome and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Principal Investigator, Angela Hillman, Assistant Professor, Ohio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18-F-13
Record Dates: First submitted 2020-06-30; First posted 2020-07-13 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Inflammation; Glucose Regulation; Sleep
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tart cherry juice concentrate (Experimental): tart cherry juice
  Interventions: Dietary Supplement: Tart cherry juice concentrate
- Freeze dried tart cherry powder (Experimental): tart cherry capsules
  Interventions: Dietary Supplement: Freeze dried tart cherry powder
- Juice placebo (Experimental): kool-aid
  Interventions: Dietary Supplement: Juice placebo
- Capsule placebo (Experimental): maltodextrin
  Interventions: Dietary Supplement: Capsule placebo

INTERVENTIONS:
Dietary Supplement: Tart cherry juice concentrate — Two 8oz bottles of tart cherry juice concentrate daily for 30 days
  Arms: Tart cherry juice concentrate
Dietary Supplement: Juice placebo — Two 8oz bottles of placebo juice daily for 30 days
  Arms: Juice placebo
Dietary Supplement: Freeze dried tart cherry powder — Two freeze dried tart cherry powder capsules daily for 30 days
  Arms: Freeze dried tart cherry powder
Dietary Supplement: Capsule placebo — Two placebo capsules daily for 30 days
  Arms: Capsule placebo

SUMMARY:
There has been a rapid increase in researching the use of tart cherry supplements in the past 5 years, particularly for inflammatory conditions. Many formulations of cherry supplements exist, however there has been no comparison between these different types. This is particularly important in the realm of inflammation research because sugar is known to increase the inflammatory response. The pill form of cherry supplementation has no added sugar and is naturally low in sugar (< 1g) while the juice form is higher from added sugar. Recent work indicates tart cherry consumption can change gut microbiota, which may modify inflammation. The purpose of this study is to look at the effects of taking a cherry supplement, either in capsule or juice form, on the gut microbiome, inflammation, and health-related variables such as blood pressure, glucose regulation and sleep quality.

DETAILED DESCRIPTION:
Participants will consume a tart cherry or placebo product for 30 days and attend 5 visits in the Exercise Physiology Lab at Ohio University over the 30 day period. They will self-collect a stool sample at baseline, 14 days and 30 days after supplementation. Blood samples will be taken at baseline, 7 days, 14 days, and 30 days after supplementation. Throughout the study participates will rate symptoms (stomach, head, etc.), pain and sleep quality using an online survey for which the link will be emailed. Participants will maintain normal diet and exercise routine and to track these for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* participate in 150 minutes of exercise per week
* non-smoker
* have no known allergy to cherries or cherry juice
* are not taking food supplements (turmeric/curcumin, cherry products, greens, etc.). -You must have access to the internet and be willing to record your food intake, physical activity and sleep quality/duration during the study.

Exclusion Criteria:

* not 18-55 years old.
* have quit smoking less than one year ago.
* have been diagnosed with a metabolic disorder such as diabetes, thyroid disorder, or high cholesterol.
* are currently being treated for arthritis or an inflammatory condition, such as arthritis, gout, lupus or Sjogren's syndrome.
* are currently being treated for cardiovascular disease, high blood pressure, fibromyalgia, or irritable bowel syndrome.
* are pregnant.
* regularly consume cherries or are allergic to cherries.
* currently use anti-inflammatory medications.
* have used corticosteroids in the last two months.
* are not willing to follow a low polyphenol diet.
* are not willing to have blood drawn on 4 occasions.
* are not willing to provide a stool sample on 3 occasions.
* do not have access to the internet.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in inflammation measured via tumor necrosis factor alpha (pg/mL) | baseline, 7 days, 14 days, and 30 days post supplementation.
Changes in inflammation measured via erythrocyte sedimentation rate (mm/hour) | baseline, 7 days, 14 days, and 30 days post supplementation.
Changes in inflammation measured via c-reactive protein (mg/L) and uric acid (mg/dL). | baseline, 7 days, 14 days, and 30 days post supplementation.
Changes in glucose regulation assessed via plasma glucose (mg/dL) | baseline, 7 days, 14 days, and 30 days post supplementation.
Changes in glucose regulation assessed via insulin (mIU/L) | baseline, 7 days, 14 days, and 30 days post supplementation.
Changes in glucose regulation assessed via glycated albumin (%). | baseline, 7 days, 14 days, and 30 days post supplementation.
Changes in sleep quantity (hours and minutes) assessed via daily survey. | daily for 30 days
Changes in sleep quality measured via 100mm visual analogue scale. | daily for 30 days
Changes in gut microbiome bacterial counts | baseline, 14 days, and 30 days post supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University Exercise Physiology Lab, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Available by request

REFERENCES:
- [Derived] Hillman AR, Chrismas BCR. Thirty Days of Montmorency Tart Cherry Supplementation Has No Effect on Gut Microbiome Composition, Inflammation, or Glycemic Control in Healthy Adults. Front Nutr. 2021 Sep 16;8:733057. doi: 10.3389/fnut.2021.733057. eCollection 2021. PMID 34604282